CLINICAL TRIAL: NCT04290065
Title: Efficacy of a Physiotherapy Intervention by Stretching the Miodural Bridge in the Modification of Posture in Professional Soccer Players. A Randomized Clinical Study.
Brief Title: Miodural Bridge Stretching in Posture Modification in Professional Footballers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Lockdown
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POST
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Hamstring Injury
Keywords: Hamstring muscle; Soccer; Flexibility; Hip joint; Suboccipital muscles
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention will take place over a period of 4 weeks, with 2 weekly sessions, with an estimated execution time of 1.50 to 3 minutes each. A manual therapy technique of inhibition of the suboccipital musculature and an axial traction of the upper hemiarchy will be performed
  Interventions: Other: Manual therapy
- Control group (No Intervention): Athletes included in the control group will not perform any intervention, continuing with their usual routine.

INTERVENTIONS:
Other: Manual therapy — The patient will be lying supine, relaxed. The physiotherapist, located at the patient's head, will cover the occipital bone with one hand while the palm of the hand will rest on the lambdoid suture, and the fingers will be introduced into the suboccipital space. The other hand, with a glove, will be inserted into the patient's oral cavity, resting respectively the index and middle fingers, each in an upper dental hemiarchy, on the chewing face of the tooth. An axial traction will be carried out until the three tension barriers of equal size between them are overcome, in an estimated time between 1.50 and 3 minutes. All manual therapy sessions will be performed by the same physiotherapist, following the same protocol and under the same conditions.
  Arms: Experimental group

SUMMARY:
Fatigue influences the kinematics of the knee. Decreasing the tone of the suboccipital musculature may decrease the tone of the knee flexors. Inhibition of the suboccipital musculature is used to improve ischiosural muscle tension.

The main objective of the study is to evaluate the effectiveness of the stretching of the miodural bridge in the modification of the posture in professional soccer players of 3rd division.

Randomized clinical trial. 30 players will be randomized to the two study groups: experimental (technique of stretching technique of the miodural bridge) and control (without intervention). A blinded evaluator will perform three evaluations: pretreatment, post-treatment and follow-up. The study variables will be: modification of posture and weight distribution (plantar pressure platform). The sample distribution will be calculated using a Kolmogórov-Smirnov analysis. The changes after each evaluation will be analyzed with the t-student test of related samples and through an ANOVA of repeated measures the intra and intersubject effect will be observed. The effect size will be calculated using Cohen's formula.

After stretching the miodural bridge, it is expected to see improvement in posture changes.

ELIGIBILITY:
Inclusion Criteria:

* Football players
* Male
* From 18 to 23 years old
* That have a federation file in 3rd division in the Region of Murcia
* That you don't have any acute lesions at the time of the study.

Exclusion Criteria:

* Subjects that: present some relevant subacute or chronic pathology that may have a direct impact on the processes or structures related to the study who have neurological problems or related to the vestibular system
* That receive a specific Physiotherapy training on any of the study regions
* Not sign the informed consent document

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline posture modification after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An evaluation will be carried out with a pedometric platform. For the evaluation of plantar pressures, we use a plantar pressure platform (Podoprint® S10Pro model). This platform has 4,096 sensors, which allow a maximum pressure of 100 N / cm2 per sensor and has a sampling frequency of 150 Hz. All measurements will be made in accordance with international standards for anthropometric evaluation. All the evaluated players will adopt a relaxed and inert bipedal orthopedic position (arms held at the sides of the body, barefoot, with clothes that allowed to see the feet, legs and knees). With eyes open and looking at a fixed point, at a distance of 1.50 m for 20 seconds.

SECONDARY OUTCOMES:
Change from baseline modification of the weight distribution after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An evaluation will be carried out with a pedometric platform, to assess the distribution of body weight after the intervention by stretching the Miodural Bridge. The unit of measure will be the percentage of weight in each of the evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain